CLINICAL TRIAL: NCT06471998
Title: Evaluation of the Benefit and Safety of Localized Tissue Hydration (HTL) in the Management of Chronic Common Low Back Pain: Phase II Monocentric Non-randomized Study
Brief Title: Evaluation of the Benefit and Safety of Localized Tissue Hydration in the Management of Chronic Low Back Pain
Acronym: HTL-LOMB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-510625-25-00
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: proof-of-concept, single-center, prospective, interventional, non-randomized Phase II study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Localized Tissue Hydration with standard care (Experimental): Localized tissue injections of saline in the routine management of pain and functional disability in patients with chronic common low back pain.
  Interventions: Drug: Sodium Chloride injection

INTERVENTIONS:
Drug: Sodium Chloride injection — Patients will receive a localized subcutaneous injection of 0.9% sodium chloride over 10 sessions (1 session per week), combined with standard treatment including stage I and II analgesics and physiotherapy in line with the recommendations of the French National Authority for Health.
  At each session, 250ml to 500ml of physiological serum will be injected subcutaneously using a Meso-Kit-Perfuser* or "injection octopus" positioned by the nurse according to the injection points defined by the investigating physician during the inclusion visit, with a dermographic tracer for surgical use.

SUMMARY:
The purpose of this study is to evaluate the benefit of Localized Tissue Hydration associated with standard management of chronic common low back pain, in terms of improvement in the numerical verbal scale score at 6 months.

DETAILED DESCRIPTION:
This is a proof-of-concept, single-center, prospective, interventional, non-randomized Phase II study designed to evaluate the benefit of 0.9% sodium chloride Localized Tissue Hydration in patients with chronic common low back pain.

The study corresponds to a clinical trial of a medicinal product in compliance with Regulation (EU) n°536/2014.

The study population is composed of patients suffering from chronic common low back pain for more than 3 months with a numerical verbal scale ≥ 5.

Patients will receive a localized subcutaneous injection of 0.9% sodium chloride over 10 sessions (1 session per week), combined with standard management including stage I and II analgesics and physiotherapy in accordance with the recommendations of the French National Authority for Health.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older ;
* Patient with chronic, non-operated low-back pain operated for more than 3 months (verbal numerical scale ≥ 5);
* Chronic common lumbago not requiring surgical management surgical ;
* Lumbar MRI performed as part of routine care and available available for the inclusion visit;
* For women of childbearing age, use of a highly effective contraceptive method;
* Patient affiliated to a French health insurance scheme;
* Patient has signed an informed consent form.

Exclusion Criteria:

* Pregnant or breast-feeding woman;
* Patient in accident at work ;
* Patient with radicular syndrome;
* Contraindication to magnetic resonance imaging or CT scan;
* Severe cases of hydric inflation and hydrosodic retention, particularly in cases of :

  * Decompensated heart failure;
  * Acute renal failure with oliguria or anuria;
  * Decompensated liver failure;
  * Pre-eclampsia/eclampsia.
* Hypochloremia ;
* Hypernatremia ;
* Patients of legal age subject to legal protection, guardianship, curatorship or deprived of liberty by judicial or administrative decision;
* Patient hospitalized without consent;
* Patient unable to answer a questionnaire;
* Patients who do not understand or speak French.

Exclusion period for inclusion in another study :

Included patients will not be allowed to participate in another interventional study during the entire follow-up period. The exclusion period is 8.5 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Success rate | 6 months
  Success rate after treatment with Localized Tissue Moisturization combined with standard management, defined by a reduction in the Verbal Numerical Scale score of at least 30%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Clairval, Marseille, France